CLINICAL TRIAL: NCT04603209
Title: Research Registry for Intra-Operative Radiotherapy (IORT) During Breast Conserving Surgery in Patients With in Situ and Early Stage Breast Cancer
Brief Title: Registry for Intra-Operative Radiotherapy During Breast Conserving Surgery in Patients With Early Stage Breast Cancer
Status: Recruiting | Type: Observational
Sponsor: Saint John's Cancer Institute (Other)
Responsible Party: Principal Investigator, Janie Grumley, Director of the Comprehensive Breast Program, Margie Petersen Breast Center, Saint John's Cancer Institute
Other Study IDs: STUDY2019000317
Record Dates: First submitted 2020-10-21; First posted 2020-10-26 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Early-stage Breast Cancer; Breast Carcinoma in Situ; Breast Neoplasms
Keywords: Breast Cancer; Early-stage Breast Cancer; Intraoperative Radiotherapy; IORT
MeSH Terms: conditions — Breast Neoplasms; Breast Carcinoma In Situ

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- IORT: All participants who plan to undergo partial mastectomy for treatment of early stage breast cancer will be considered for eligibility for IORT. Patient with single breast cancer less than 3cm in disease span, clinical negative axillary node will be offered the option of having IORT. If IORT is delivered following surgical resection of the tumor they will be followed in this registry for short and long term outcomes.
  Interventions: Radiation: Intraoperative Radiation Therapy (IORT)

INTERVENTIONS:
Radiation: Intraoperative Radiation Therapy (IORT) — IORT involving 50kV Xrays to a dose of 20 Gy during breast-conserving surgery

SUMMARY:
This is a prospective, registry study that will enroll all women with early stage breast cancer who will be treated with intraoperative radiotherapy (IORT) during breast-conserving surgery. The purpose of this study is to further validate the long-term effectiveness and safety of this treatment method. We aim to assess short and long-term patient outcomes associated with IORT, including perioperative complications, local and distance disease recurrences, as well as disease-free survival and overall survival.

DETAILED DESCRIPTION:
At Providence Saint John's Health Center, there is the ongoing integration of Intra-Operative Radiation Therapy (IORT) as a standard treatment option among Breast Conserving Therapy (BCT) for individuals with in situ and early stage breast cancer. Currently, approximately 60 women per year are being treated with IORT. No repository of information of patient outcomes with this treatment has been established. This leaves a critical gap in the ability to assess the long-term outcomes of patients treated with IORT.

As the practice of using IORT to treat early stage and in situ breast cancer continues to grow at Providence Saint John's Health Center, this registry will provide the data needed to compare patient outcomes with those being treated with the traditional whole breast radiation therapy. In addition, the Providence Health & Services strives to improve patient care and outcomes with excellence whenever possible. The registry will provide the data needed to compare patient outcomes to national and community standards that can inform internal practice patterns and contribute to advancing breast cancer care nationally and internationally.

ELIGIBILITY:
Inclusion Criteria:

* Clinical stage Tis, T1, or T2(≤ 3cm), N0, M0 (AJCC Classification)
* Unifocal Disease
* Candidate for breast-conserving surgery
* Recommended treatment by multidisciplinary team

Exclusion Criteria:

* Clinical stage T3-4, N1-3, M1
* Multifocal disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any individual aged ≥ 18 years with early stage breast cancer who is determined to be suitable candidates for breast-conserving surgery and IORT by a multidisciplinary team.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2018-10-03 (Actual); Primary Completion 2028-10-03 (Estimated); Study Completion 2028-10-03 (Estimated)

PRIMARY OUTCOMES:
Disease Recurrence | 5 years
  Presence of recurrent tumor in ipsilateral breast or distant site

SECONDARY OUTCOMES:
Disease specific survival | 10 years
  survival
Overall Survival | 10 years
  survival

CONTACTS AND LOCATIONS:
Overall Officials: Janie Grumley, MD, Principal Investigator — John Wayne Cancer Institute, Providence Saint John's Health Center
Locations (1):
- John Wayne Cancer Institute, Providence Saint John's Health Center, Santa Monica, California, United States